CLINICAL TRIAL: NCT06939348
Title: Safety and Efficacy of Thalamic Focused Ultrasound Stimulation (tFUS) for Promoting Recovery After Severe Traumatic Brain Injury
Brief Title: Ultrasound Stimulation for Patients in a Disorder of Consciousness
Acronym: tFUS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: Casa Colina Hospital and Centers for Healthcare (Other); Spaulding Rehabilitation Hospital (Other); Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Martin M Monti, Associate Professor, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB-24-1241; TP230324 (Other Grant/Funding Number: US Department of Defense-Traumatic Brain Injury and Psychological Health Research Program--Clinical Trial Award (RL2))
Record Dates: First submitted 2025-04-07; First posted 2025-04-22 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2025-04

CONDITIONS: Consciousness Disorders; Disorders of Consciousness Due to Severe Brain Injury
Keywords: Disorder of Consciousness; Vegetative State; Minimally Conscious State; Minimally Conscious State Plus; Minimally Conscious State Minus; Traumatic Brain Injury; CVA (Cerebrovascular Accident); Anoxia, Brain; Thalamic Infarction; Coma; Prolonged
MeSH Terms: conditions — Consciousness Disorders; Persistent Vegetative State; Brain Injuries, Traumatic; Stroke; Hypoxia, Brain; Coma

STUDY DESIGN:
Intervention Model Description: Sham-controlled 2-arm design. The clinical trial study features a 2-arm, sham-controlled, design. One group will be randomized to receive pulsed thalamic tFUS. The second group will undergo sham procedure. The sham procedure is identical to previous tFUS procedure (NCT04921683), except the gel pad used to couple the transducer to the patient's head is "non-transmitting" (as opposed to "transmitting"), thus preventing any penetration of ultrasound inside the head.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Sham-tFUS group (Sham Comparator): Sham-tFUS group will receive sham sonication in the first session and tFUS in the second session
  Interventions: Device: The Brainsonix BX Pulsar 1002 was designed to deliver low-intensity focused ultrasound pulsations (LIFUP) to the human brain.
- tFUS-tFUS group (Active Comparator): tFUS-tFUS group will receive 2 sessions of tFUS
  Interventions: Device: The Brainsonix BX Pulsar 1002 was designed to deliver low-intensity focused ultrasound pulsations (LIFUP) to the human brain.

INTERVENTIONS:
Device: The Brainsonix BX Pulsar 1002 was designed to deliver low-intensity focused ultrasound pulsations (LIFUP) to the human brain. — The BX Pulsar 1002 consists of two main elements: the transducer and the ultrasound console. The transducer itself and the housing for it went through several iterations in order to be compatible with an MRI environment. Currently, the transducer and its housing are deemed MR-conditional at 3T with SAR ≤ 2W/kg. The design includes a solid acoustic coupling gel pad attached to the front of the transducer to provide good acoustic transmission into the scalp. An outer housing was designed to attach the transducer firmly to the head above the temporal window, and to allow it to be moved side to side to accurately target intended structures.

SUMMARY:
The overall aim of this study is to develop an intervention that can help recovery in patients surviving severe brain injury but failing to fully recover. In particular, this multicenter project aims to (1) establish short-term efficacy of tFUS as a therapeutic to promote recovery in patients with prolonged DoC as compared to sham treatment, (2) establish dose-related safety and efficacy of tFUS as a therapeutic intervention in prolonged DoC patients and (3) explore preliminary predictors and biomarkers of susceptibility and response to thalamic sonication.

DETAILED DESCRIPTION:
Aim 1 - Establish short-term efficacy of tFUS as a therapeutic to promote recovery in patients with prolonged DoC as compared to sham treatment. Investigators will use a multicenter sham-controlled randomized double-blind design to test the efficacy of tFUS for the recovery of consciousness in prolonged DoC, secondary to TBI. Specifically, The investigators will use a sham that is identical to a previous procedure (NCT04921683), except the gel pad used to couple the transducer to the patient's head is "non-transmitting" (as opposed to "transmitting"), thus preventing any penetration of ultrasound inside the head. Approach overview: 40 patients in a prolonged DoC due to TBI (> 28days post injury) will be randomized into one of two conditions: (a) the tFUS-tFUS group will receive 2 sessions of tFUS and (b) the Sham-tFUS group will receive sham sonication in the first session and tFUS in the second session. Measurements: Outcome measures collected prior to tFUS/sham sessions will be compared to outcome measures obtained one week after tFUS/sham sessions. The investigators will assess two endpoint measures: one DoC-specific (i.e., the Coma Recovery Scale Revised - CRS-R; primary measure) [17] (Aim 1a) and one specific to TBI functional outcome (i.e., the Disability Rating Scale; secondary measure) [18] (Aim 1b). Hypotheses Compared to the sham condition, tFUS will lead to a statistically significant increase in consciousness recovery (Aim 1a) and in functional recovery (Aim 1b).

Aim 2 - Establish dose-related safety and efficacy of tFUS as a therapeutic intervention in prolonged DoC patients. Approach overview: The investigators will assess and compare safety and efficacy data in both conditions (ie, the tFUS-tFUS group who will receive 2 tFUS sessions and the Sham-tFUS group who will receive one tFUS session). Measurements: Safety. Proportion of (severe) adverse events (primary measure) will be documented using the Adverse Event Questionnaire (AEQ, also used in NCT04921683) and the Vital signs Care Report Form (CRF) (Common Data Element F0026), [6] within one week of intervention/sham, in the tFUS-tFUS group and in the Sham-tFUS group (Aim 2a); Efficacy. Changes will be assessed, one week after intervention/sham, in the tFUS-tFUS group as compared to the Sham-tFUS group using the CRS-R (secondary measure) (Aim 2b). Hypotheses: Aim 2a: Applying 2 sessions of tFUS will not lead to (higher proportion of) adverse events; Aim 2b: A statistically significant increase in consciousness recovery will be observed when applying two versus one tFUS sessions.

Aim 3 - Explore preliminary predictors and biomarkers of susceptibility and response to thalamic sonication. The investigators will assess pre-post intervention-related changes in brain activity using electrophysiology in both conditions (i.e., tFUS-tFUS group vs. Sham-tFUS group) (Aim 3a). The investigators will also assess whether the effects of tFUS are TBI-specific by comparing the efficacy observed in our TBI group vs. a non-TBI group (Aim 3b). Approach overview: In addition to our two endpoint measures (i.e., DRS and CRS-R), a 15-minute resting electroencephalogram (EEG) will be collected immediately before and after each tFUS or sham session (Aim 3a). Efficacy (as described in Aim 1a) will be additionally tested in 20 patients in a prolonged DoC due to non-TBI causes (> 28days post injury due to stroke or anoxia) to help determine if tFUS is a TBI specific treatment (Aim 3b). Measurements: For Aim 3a, using the EEG recordings, power spectral density will be calculated within predefined frequency band and ABCD level classification (that reflects the degree of thalamocortical disconnection; primary measure) [7] will be applied based on spectral peaks in these frequencies. For Aim 3b, TBI specific efficacy will be tested based on the change observed one week after tFUS sessions as compared to sham sessions using the CRS-R (secondary measure) in both TBI and non-TBI groups. Hypothesis: Aim 3a: tFUS, but not sham will promote recovery of thalamocortical integrity as estimated by the ABCD level classification based on the Mesocircuit theory [2]; Aim 3b: Compared to sham, tFUS will lead to a statistically significant increase in consciousness recovery, particularly, in the TBI group vs. the non-TBI group.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of DoC, following international guidelines, as assessed with the CRS-R.
2. Prolonged status (>28days post-injury)
3. If on a psychotropic medication regimen, that regimen will be stable for at least 4 weeks prior to entry to the study and the patient will be willing to remain on a stable regimen during the protocol.
4. legally authorized representative available to consent for the patient to participate in the study

Exclusion Criteria:

1. History of neurological disorder (other than the brain injury).
2. Metal implant or other condition precluding safe entry in the MR-environment.
3. Manifest continuous spontaneous movement (which would prevent safe/successful imaging).
4. Participation in another concurrent clinical trial.
5. Need for mechanical ventilation.
6. Craniotomy (no bone flap).
7. Cranioplasty spanning the left temporal bone window.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-04-26 (Actual); Primary Completion 2028-03-28 (Estimated); Study Completion 2028-09-29 (Estimated)

PRIMARY OUTCOMES:
Establish short-term efficacy of tFUS as a therapeutic to promote recovery in patients with prolonged DoC as compared to sham treatment. | From Day 1 to 16
  Outcome measures collected prior to tFUS/sham sessions will be compared to outcome measures obtained one week after tFUS/sham sessions. The two endpoint measures used will be one DoC-specific measure: the Coma Recovery Scale Revised (CRS-R). The Coma Recovery Scale Revised (CRS-R) ranges from 0 to 23 points, with higher scores indicating better neurological function and level of consciousness. A score of 0 represents the lowest level of neurological functioning, while a score of 23 represents the highest level of neurological functioning.
Establish dose-related safety and efficacy of tFUS as a therapeutic intervention in prolonged DoC patients. | From Day 1 to 16
  Safety. Proportion of (severe) adverse events (primary measure) will be documented using the Adverse Event Questionnaire (AEQ, also used in NCT04921683) and the Vital signs CRF (F0026),22 within one week of intervention/sham, in the tFUS-tFUS group and in the Sham-tFUS group
Explore preliminary predictors and biomarkers of susceptibility and response to thalamic sonication. | From Day 1 to 16
  using the EEG recordings, power spectral density will be calculated within predefined frequency band and ABCD level classification (that reflects the degree of thalamocortical disconnection; primary measure) will be applied based on spectral peaks in these frequencies. This measure is calculated in percentage (%) of total power density.

SECONDARY OUTCOMES:
Establish short-term efficacy of tFUS as a therapeutic to promote recovery in patients with prolonged DoC as compared to sham treatment | From Day 1 to 16
  Outcome measures collected prior to tFUS/sham sessions will be compared to outcome measures obtained one week after tFUS/sham sessions. The two endpoint measures used will be one specific to TBI functional outcome: the Disability Rating Scale (DRS). The Disability Rating Scale (DRS) ranges from 0 to 30 points, with higher scores indicating more severe disability. A score of 0 represents no disability, while a score of 30 represents extreme vegetative state or death.
Establish dose-related safety and efficacy of tFUS as a therapeutic intervention in prolonged DoC patients. | From Day 1 to 16
  Efficacy. Changes will be assessed, one week after intervention/sham, in the tFUS-tFUS group as compared to the Sham-tFUS group using the CRS-R. The Coma Recovery Scale Revised (CRS-R) ranges from 0 to 23 points, with higher scores indicating better neurological function and level of consciousness. A score of 0 represents the lowest level of neurological functioning, while a score of 23 represents the highest level of neurological functioning.
Explore preliminary predictors and biomarkers of susceptibility and response to thalamic sonication. | From Day 1 to 16
  TBI specific efficacy will be tested based on the change observed one week after tFUS sessions as compared to sham sessions using the CRS-R (secondary measure) in both TBI and non-TBI groups

CONTACTS AND LOCATIONS:
Overall Officials: Martin M Monti, PhD, Principal Investigator — University of California, Los Angeles
Locations (4):
- United States (4):
  - The Regents of the University of California, Los Angeles, Los Angeles, California
  - Casa Colina Hospital and Centers for Healthcare, Pomona, California
  - Massachusetts General Hospital (The General Hospital Corp.), Boston, Massachusetts
  - Spaulding Rehabilitation Hospital Corporation, Inc., Charlestown, Massachusetts

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lutkenhoff ES, Chiang J, Tshibanda L, Kamau E, Kirsch M, Pickard JD, Laureys S, Owen AM, Monti MM. Thalamic and extrathalamic mechanisms of consciousness after severe brain injury. Ann Neurol. 2015 Jul;78(1):68-76. doi: 10.1002/ana.24423. Epub 2015 May 4. PMID 25893530
- [Result] Sanz LRD, Lejeune N, Blandiaux S, Bonin E, Thibaut A, Stender J, Farber NM, Zafonte RD, Schiff ND, Laureys S, Gosseries O. Treating Disorders of Consciousness With Apomorphine: Protocol for a Double-Blind Randomized Controlled Trial Using Multimodal Assessments. Front Neurol. 2019 Mar 19;10:248. doi: 10.3389/fneur.2019.00248. eCollection 2019. PMID 30941094
- [Result] Bogner JA, Whiteneck GG, MacDonald J, Juengst SB, Brown AW, Philippus AM, Marwitz JH, Lengenfelder J, Mellick D, Arenth P, Corrigan JD. Test-Retest Reliability of Traumatic Brain Injury Outcome Measures: A Traumatic Brain Injury Model Systems Study. J Head Trauma Rehabil. 2017 Sep/Oct;32(5):E1-E16. doi: 10.1097/HTR.0000000000000291. PMID 28195954
- [Result] Thibaut A, Bruno MA, Ledoux D, Demertzi A, Laureys S. tDCS in patients with disorders of consciousness: sham-controlled randomized double-blind study. Neurology. 2014 Apr 1;82(13):1112-8. doi: 10.1212/WNL.0000000000000260. Epub 2014 Feb 26. PMID 24574549
- [Result] Kalmar K, Giacino JT. The JFK Coma Recovery Scale--Revised. Neuropsychol Rehabil. 2005 Jul-Sep;15(3-4):454-60. doi: 10.1080/09602010443000425. PMID 16350986
- [Result] Schnakers C, Monti MM. Disorders of consciousness after severe brain injury: therapeutic options. Curr Opin Neurol. 2017 Dec;30(6):573-579. doi: 10.1097/WCO.0000000000000495. PMID 28901969
- [Result] Gosseries O, Demertzi A, Ledoux D, Bruno MA, Vanhaudenhuyse A, Thibaut A, Laureys S, Schnakers C. Burnout in healthcare workers managing chronic patients with disorders of consciousness. Brain Inj. 2012;26(12):1493-9. doi: 10.3109/02699052.2012.695426. Epub 2012 Jun 22. PMID 22725684
- [Result] Jennett B. Thirty years of the vegetative state: clinical, ethical and legal problems. Prog Brain Res. 2005;150:537-43. doi: 10.1016/S0079-6123(05)50037-2. PMID 16186047
- [Result] Monti MM, Laureys S, Owen AM. The vegetative state. BMJ. 2010 Aug 2;341:c3765. doi: 10.1136/bmj.c3765. No abstract available. PMID 20679291
- [Result] Monti MM. Cognition in the vegetative state. Annu Rev Clin Psychol. 2012;8:431-54. doi: 10.1146/annurev-clinpsy-032511-143050. Epub 2012 Jan 3. PMID 22224835
- [Result] Tufail Y, Yoshihiro A, Pati S, Li MM, Tyler WJ. Ultrasonic neuromodulation by brain stimulation with transcranial ultrasound. Nat Protoc. 2011 Sep 1;6(9):1453-70. doi: 10.1038/nprot.2011.371. PMID 21886108
- [Result] Folloni D, Verhagen L, Mars RB, Fouragnan E, Constans C, Aubry JF, Rushworth MFS, Sallet J. Manipulation of Subcortical and Deep Cortical Activity in the Primate Brain Using Transcranial Focused Ultrasound Stimulation. Neuron. 2019 Mar 20;101(6):1109-1116.e5. doi: 10.1016/j.neuron.2019.01.019. Epub 2019 Feb 11. PMID 30765166
- [Result] Yoo SS, Kim H, Min BK, Franck E, Park S. Transcranial focused ultrasound to the thalamus alters anesthesia time in rats. Neuroreport. 2011 Oct 26;22(15):783-7. doi: 10.1097/WNR.0b013e32834b2957. PMID 21876461
- [Result] Deffieux T, Younan Y, Wattiez N, Tanter M, Pouget P, Aubry JF. Low-intensity focused ultrasound modulates monkey visuomotor behavior. Curr Biol. 2013 Dec 2;23(23):2430-3. doi: 10.1016/j.cub.2013.10.029. Epub 2013 Nov 14. PMID 24239121
- [Result] Legon W, Sato TF, Opitz A, Mueller J, Barbour A, Williams A, Tyler WJ. Transcranial focused ultrasound modulates the activity of primary somatosensory cortex in humans. Nat Neurosci. 2014 Feb;17(2):322-9. doi: 10.1038/nn.3620. Epub 2014 Jan 12. PMID 24413698
- [Result] Bystritsky A, Korb AS, Douglas PK, Cohen MS, Melega WP, Mulgaonkar AP, DeSalles A, Min BK, Yoo SS. A review of low-intensity focused ultrasound pulsation. Brain Stimul. 2011 Jul;4(3):125-36. doi: 10.1016/j.brs.2011.03.007. Epub 2011 Apr 1. PMID 21777872
- [Result] Monti MM, Schnakers C, Korb AS, Bystritsky A, Vespa PM. Non-Invasive Ultrasonic Thalamic Stimulation in Disorders of Consciousness after Severe Brain Injury: A First-in-Man Report. Brain Stimul. 2016 Nov-Dec;9(6):940-941. doi: 10.1016/j.brs.2016.07.008. Epub 2016 Jul 22. No abstract available. PMID 27567470
- [Result] Tsubokawa T, Yamamoto T, Katayama Y, Hirayama T, Maejima S, Moriya T. Deep-brain stimulation in a persistent vegetative state: follow-up results and criteria for selection of candidates. Brain Inj. 1990 Oct-Dec;4(4):315-27. doi: 10.3109/02699059009026185. PMID 2252964
- [Result] Schiff ND, Giacino JT, Kalmar K, Victor JD, Baker K, Gerber M, Fritz B, Eisenberg B, Biondi T, O'Connor J, Kobylarz EJ, Farris S, Machado A, McCagg C, Plum F, Fins JJ, Rezai AR. Behavioural improvements with thalamic stimulation after severe traumatic brain injury. Nature. 2007 Aug 2;448(7153):600-3. doi: 10.1038/nature06041. PMID 17671503
- [Result] Schiff ND. Recovery of consciousness after brain injury: a mesocircuit hypothesis. Trends Neurosci. 2010 Jan;33(1):1-9. doi: 10.1016/j.tins.2009.11.002. Epub 2009 Dec 1. PMID 19954851
- [Result] Monti MM, Rosenberg M, Finoia P, Kamau E, Pickard JD, Owen AM. Thalamo-frontal connectivity mediates top-down cognitive functions in disorders of consciousness. Neurology. 2015 Jan 13;84(2):167-73. doi: 10.1212/WNL.0000000000001123. Epub 2014 Dec 5. PMID 25480912
- [Result] Lutkenhoff ES, McArthur DL, Hua X, Thompson PM, Vespa PM, Monti MM. Thalamic atrophy in antero-medial and dorsal nuclei correlates with six-month outcome after severe brain injury. Neuroimage Clin. 2013 Oct 5;3:396-404. doi: 10.1016/j.nicl.2013.09.010. eCollection 2013. PMID 24273723